CLINICAL TRIAL: NCT06826365
Title: Analysis of Immune Cell Populations in the Endometrium and Peripheral Blood in Women With Reduced and Normal Fertility
Brief Title: Immune Cell Populations in the Endometrium
Status: Not yet recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, PhD, MD, Principal Investigator, Jagiellonian University
Other Study IDs: 1072.6120.301.2022
Record Dates: First submitted 2025-02-08; First posted 2025-02-14 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Infertility, Female; Recurrent Miscarriage; Gynecologic Disease
Keywords: Idiopathic infertility; Endometrial immunology; Endometrial aspiration biopsy; Recurrent miscarriage
MeSH Terms: conditions — Infertility, Female; Abortion, Habitual; Genital Diseases, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * 1 ml endometrial sample
  * 10 ml peripheral blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infertility: Women aged 18-45 with idiopathic infertility/recurrent miscarriages
  Interventions: Diagnostic Test: Percentage distribution of immune system cells in peripheral blood; Diagnostic Test: Percentage distribution of immune system cells in endometrium
- Normal fertility: Women aged 18-45 with a history of normal pregnancy obtained by spontaneous fertilization
  Interventions: Diagnostic Test: Percentage distribution of immune system cells in peripheral blood; Diagnostic Test: Percentage distribution of immune system cells in endometrium

INTERVENTIONS:
Diagnostic Test: Percentage distribution of immune system cells in peripheral blood — Assessment of the percentage distribution of the immune system cell population in peripheral blood by flow cytometry
Diagnostic Test: Percentage distribution of immune system cells in endometrium — Assessment of the percentage distribution of the immune system cell population in endometrium by flow cytometry

SUMMARY:
Specialized immunological studies in the diagnostics of idiopathic infertility and recurrent miscarriages have limited applicability, as the role of the immune system in these conditions is not thoroughly understood. In ovulatory cycles, changes occur in the populations of uterine lymphocytes, which may influence the receptivity of the endometrium and the implantation of the embryo. Particularly notable are the changes in natural killer (NK) cells, which reach their peak during the luteal phase and regulate the invasion of the trophoblast. The dominant NK cells exhibit a CD56bright phenotype and differ in cytokine profiles from peripheral blood cells. Cyclical changes also affect macrophages and T lymphocytes; however, it is unclear whether their proportions differ in women with reduced fertility. There is a need to investigate how the composition of lymphocytes in blood influences the populations in the endometrium. The aim of this study is to analyze the correlation between peripheral and endometrial lymphocytes in women with idiopathic infertility and recurrent miscarriages, compared to fertile women.

DETAILED DESCRIPTION:
A cross-sectional study will be conducted among women aged 18-45 years undergoing aspiration biopsy as part of the diagnosis of: i) idiopathic infertility, ii) recurrent miscarriages, iii) other conditions requiring histopathological examination of the endometrium (control).

A 2 ml endometrial biopsy will be collected using the NEXODIS suction cannula on day 20-22 of the cycle, after confirmation of a negative result of B-human chorionic gonadotropin in the blood, and divided into 2 parts: 1 ml will be secured and sent for cytometric examination. At the same time, a peripheral blood sample (10 ml) will be collected in accordance with the SU in-hospital procedure and sent for cytometric examination.

Labeled blood cells and isolated single endometrial cells will be analyzed by flow cytometry using the FACSCanto2 system (BD Biosciences, USA). Blood cells will be stained directly with a panel of antibodies, and endometrial samples will be crushed and filtered before staining to isolate single cells. Then, the stained cells will be washed, erythrocytes will be lysed and centrifuged. It is planned to use a panel of monoclonal antibodies conjugated with fluorochromes, recognising the following markers: CD45, CD56, CD16, CD3, CD64, CD206, CD163, CD80, CD86 and CD138. The study population will be characterised in terms of age, BMI, gynecological data (surgeries, course of the menstrual cycle, nature of bleeding, ultrasound data) and obstetric data (pregnancies, deliveries, miscarriages). Characteristics of the study population, results of cytometric, histopathological, immunohistochemical endometrial and blood cytometric tests and their mutual correlation will be analysed using standard statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years
* idiopathic infertility
* at least 2 miscarriages
* other benign gynecological conditions subjected to endometrial sampling

Exclusion Criteria:

* miscarriage within last 3 months
* abdominal/uterine surgery within last 3 months
* viral/bacterial infection within last 3 months
* antibiotic therapy within last 3 months

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women undergoing endometrial aspiration biopsy for the diagnosis of: i) idiopathic infertility, ii) recurrent miscarriages, iii) other conditions requiring histopathological examination of the endometrium (control).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the percentage of Non-classical monocytes CD16++/ CD14- (% monocytes) in peripheral blood | up to 6 months
  Comparison of the percentage of Non-classical monocytes CD16++/ CD14- (% monocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of Intermediate monocytes CD16+/CD14+ (% monocytes) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of Intermediate monocytes CD16+/CD14+ (% monocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of Classical monocytes CD16-/CD14++ (% monocytes) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of Classical monocytes CD16-/CD14++ (% monocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of plasmocytes (% leukocytes) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of plasmocytes (% leukocytes) in both study arms - in the group with normal and reduced fertility
Assessment of Macrophages M1/M2 CD163+/CD206- (% monocytoid cells) ratio in peripheral blood | up to 6 months
  Comparison of the Macrophages M1/M2 CD163+/CD206- (% monocytoid cells) ratio in peripheral blood in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of CD3+ lymphocytes (% lymphocytes) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of CD3+ lymphocytes (% lymphocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of B lymphocytes (% lymphocytes) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of B lymphocytes (% lymphocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of Total NK (% lymphocytes) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of Total NK (% lymphocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of NK CD56++/CD16- (% NK) in peripheral blood | up to 6 months
  Comparison of the percentage of NK CD56++/CD16- (% NK) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of NK CD56+/CD16+ (% NK) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56+/CD16+ (% NK) in both study arms - in the group with normal and reduced fertility fertility
Assessment of the percentage of NK CD56+/CD16++ (% NK) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56+/CD16++ (% NK) in both arms of the study - in the group with normal and reduced fertility
Assessment of the percentage of NK CD56-/CD16++ (% NK) in peripheral blood by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56-/CD16++ (% NK) in both arms of the study - in the group with normal and reduced fertility
Assessment of the percentage of Non-classical monocytes CD16++/ CD14- (% monocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of Non-classical monocytes CD16++/ CD14- (% monocytes) in both study arms - in the group with normal and reduced fertility
ssessment of the percentage of Intermediate monocytes CD16+/CD14+ (% monocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of Intermediate monocytes CD16+/CD14+ (% monocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of Classical monocytes CD16-/CD14++ (% monocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of Classical monocytes CD16-/CD14++ (% monocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the ratio of Macrophages M1/M2 CD163+/CD206- (% monocytoid cells) in endometrium by flow cytometry | up to 6 months
  Comparison of the ratio of Macrophages M1/M2 CD163+/CD206- (% monocytoid cells) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of plasmocytes (% leukocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of plasmocytes (% leukocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of CD3+ lymphocytes (% lymphocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of CD3+ lymphocytes (% lymphocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of B lymphocytes (% lymphocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of B lymphocytes (% lymphocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of Total NK (% lymphocytes) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of Total NK (% lymphocytes) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of NK CD56++/CD16- (% NK) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56++/CD16- (% NK) in both study arms - in the group with normal and reduced fertility
Assessment of the percentage of NK CD56+/CD16+ (% NK) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56+/CD16+ (% NK) in both study arms - in the group with normal and reduced fertility fertility
Assessment of the percentage of NK CD56+/CD16++ (% NK) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56+/CD16++ (% NK) in both arms of the study - in the group with normal and reduced fertility
Assessment of the percentage of NK CD56-/CD16++ (% NK) in endometrium by flow cytometry | up to 6 months
  Comparison of the percentage of NK CD56-/CD16++ (% NK) in both arms of the study - in the group with normal and reduced fertility

CONTACTS AND LOCATIONS:
Overall Officials: Kazimierz Pityński, Prof., PhD, Study Chair — Jagiellonian University